CLINICAL TRIAL: NCT02718612
Title: Association Between Sarcopenia and Sarcopenic Obesity With Metabolic and Cardiovascular Risk Factors in Taiwanese Dialysis Patients
Brief Title: Prevalence and Determinants of Sarcopenic Obesity in Taiwanese Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Principal Investigator, Paik Seong Lim, MD, Tungs' Taichung Metroharbour Hospital
Other Study IDs: 104079
Record Dates: First submitted 2016-03-04; First posted 2016-03-24 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Sarcopenia
Keywords: Uraemic Sarcopenia; Sarcopenic Obesity
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Uraemic sarcopenia is complex, and progressive . As older persons are particularly susceptible to renal failure and this accelerates the physiological muscle wasting in this patient group. Hence sarcopenia is an important factor of functional impairment in elderly patients suffering from chronic kidney disease. On the other hand, overweight has become increasing common in dialysis patients, and is paradoxically reported to be associated with better survival. It remains unclear if adipose tissue in overweight in elderly dialysis patients is a source of proinflammatory mediators, which could contribute to protein-energy wasting (PEW), cardiovascular disease, and increased mortality. This study attempts to explore the prevalence of Sarcopenic Obesity (SO) in a cohort of hemodialysis patients with a more well defined criteria. In addition, this study aims to examine the association between sarcopenia and SO with metabolic and cardiovascular risk factors in these patients.

DETAILED DESCRIPTION:
Patients

The study is a cross-sectional analysis of all patients on hemodialysis patients treated at Tungs' Taichung Metroharbor hospital(500 patients). Patients ≥20 years of age and been on maintenance hemodialysis for at least 3 month before the study. The dialysis sessions were 3.5 to 4.5 h three times per week, with a blood flow greater than 300 mL/min, a dialysate flow of 600 mL/min, and a bicarbonate buffer.

Clinical assessments and data collection

The investigators collect baseline clinical data [such as age, sex, height, bodyweight, clinical etiology of Chronic Kidney Disease if possible, comorbidities, blood pressure, laboratory measures [such as serum creatinine, albumin, C-reactive protein (CRP), total cholesterol, complete blood counts, total carbon dioxide, anthropometric information and various potential indicators of PEW [such as body mass index, waist/hip ratio, mid-arm circumference (MAC), triceps skinfold thickness (TSF), mid-arm muscle circumference (MAMC), mid-arm muscle area (MAMA), SGA, BIA analyses, and hand grip Strength (HGS). For the laboratory tests, fasting blood samples are obtained from each patient and are performed in the Department of Clinical Pathology of the investigators hospital by means of routine methods. Interleukin-6 (IL-6) and tumour necrosis factor-α(TNF-α )levels are measured via immunometric enzyme immunoassay. Insulin is analyzed using human ELISA kits . Sensitivity is 2.88 pmol/L, and the upper limits of intra- and inter-assay coefficients of variation were 3.3 and 7.6, respectively. Homeostatic Model Assessment Insulin Resistance(HOMA-IR) was calculated as fasting insulin (U/l) × fasting glucose (mg/dl)/405, as described by Matthews et al.

All patients received echocardiograms studies performed within 3 months after enrollment, which were used to estimate Congestive Heart Failure (defined as an ejection fraction of <40%) or left ventricular hypertrophy (LVH, defined as left ventricle mass index 125 g/m2 in men and 100 g/m2 in women). Cardiovascular disease is defined as a previous history of Congestive Heart Failure, LVH, ischemic heart disease(including prior history of angina, myocardial infarction, coronary artery bypass grafting and percutaneous cardiac catheter intervention) or cerebrovascular disease (including prior history of transient ischemic attack and stroke).

Anthropometric measurements

The actual bodyweight and height on the day of assessment was used. Anthropometric measurements include TSF used skinfold calipers MAC measured by a stretchable measuring tape, MAMC equals MAC(centimeter) -3.14 x TSF (millimeter)/10 and MAMA equals (MAMC2/4π).

Body composition measurements

1. Bioelectrical impedance analysis (BIA) device :(Tanita BC-418) Body composition was measured using an 8-contact electrode bioelectrical impedance analysis (BIA) device (Tanita BC-418, Tanita, Tokyo, Japan), as well as BIS (FMC) and followed the standard procedure and the manufacturer's instructions.This BIA device was used to measure the whole body and segmental impedance (± 1Ω) at a frequency of 50 kilohertz (kHz), and it provided valid muscle mass estimates (kg) of each of the four extremities. Appendicular muscle mass (ASM) was calculated as the sum of the estimated muscle mass for the arms and legs. A relative skeletal muscle mass index (ASM/ht2) normalized for height was defined as the ratio of ASM (kg) and the height squared(m2). For this analysis, the investigators defined muscle mass cut-off points according to the distribution of ASM/ht2 of a young population comprising 998 healthy adults (aged 20-40 years) or the study population. A participant was considered to have low muscle mass if his or her ASM/ht2 was below -2 standard deviations of the reference young adult values defined in previous studies (6.76 kg/m2 for men and 5.28 kg/m2 for women).
2. Bioelectric impedance spectroscopy (BIS)

BIS measurement was performed in each of the participants enrolled in the study by a specific member of staff who had completed a training course in the BIS technique, using a portable whole body bioimpedance spectroscopy device, the body composition monitor (BCM: Fresenius Medical Care, Bad Homburg, Germany). The BCM measures the impedance spectroscopy at 50 different frequencies between 5 kHz and 1 megahertz (MHz). Measurements were taken on the midweek dialysis session before the start of the hemodialysis treatment with the patient calm, supine, and relaxed in the dialysis bed for 10 minutes. Specific exclusion criteria were dictated by the device and included history of a pacemaker, defibrillator, metallic sutures, or stent implantation and amputation of a major limb. The device expresses the body weight in terms of lean tissue mass (LTM - mainly muscle), adipose tissue mass (ATM - mainly fat) and overhydration(OH). Each of these compartments has a specific composition and contains a known quantity of water per mass of tissue. Overhydration(OH) is almost 100% extracellular water, whereas the water of LTM and ATM consist of differing proportion of extracellular and intracellular water in addition to solid components.

Gait speed

Participants were observed taking a walk over a short distance at their usual pace, starting from a standing position, and an examiner timed the task by using a handheld stopwatch that measured to the nearest hundredth of a second. The walking distance ranged from 3 to 5 m according to different study sites. The gait speed was calculated as the walking distance (m) divided by time (s). The investigators examined the distribution of the gait speed stratified according to the sex-specific median height. Participants with a gait speed in the lowest 20% of the sex- and height-specific distributions were considered to have low gait speed.

Handgrip strength

Handgrip strength is measured on the non-fistula side before a dialysis session using mechanical dynamometers with a precision of less than 0.5 kg. Subjects are instructed to self-adjust the dynamometer so that it fit comfortably to their hand size to obtain the best performance. Before data collection, a warm up section is conducted so that the subjects could become acquainted with the instrument and procedures and choose the best adjustment. Subjects are instructed to grip the dynamometer with maximum strength in response to a voice command. The subjects stand with both arms extended sideways from the body with the dynamometer facing away from the body. Three trials are performed with a rest period of at least 1 min between trials and the highest HGS value is used in the analyses. Participants with a handgrip strength in the lowest 20% of the sex- and BMI-specific distributions are considered to have low handgrip strength.

Assessments of nutritional status and potential indicators of PEW

Subjective Global Assessment (SGA)

The SGA is recommended by National Kidney Foundation Kidney / Disease Outcomes Quality Initiative(K/DOQI) as an instrument for assessing the nutritional status of dialysis patients . It is a semiquantitative scoring system based on history and physical examination. The history consists of five components: weight loss during the preceding 6 months, gastrointestinal symptoms, food intake, functional capacity, and comorbidities. Each of these features is scored separately as A, B, or C, reflecting well-nourished to severely malnourished categories. The physical examination consists of 2 components: loss of subcutaneous fat and muscle wasting. These two components are classified in terms of the three major SGA scores: A, well nourished; B, mild to moderate malnutrition; and C, severe malnutrition.

Malnutrition-Inflammation Score (MIS)

MIS scoring sheet consists of four sections (patient's related medical history, physical examination, body mass index (BMI), and laboratory parameters) and 10 components. Patient's medical history consists of five components: dry weight changes, dietary intake, gastrointestinal symptoms, functional capacity, and co-morbidity, including number of years on dialysis. Major comorbid conditions (MCC) include congestive heart failure class III or IV, , severe coronary artery disease, moderate to severe chronic obstructive pulmonary disease (COPD), major neurological sequelae, and metastatic malignancies or status post recent chemotherapy. Physical examination consists of two components, which aims to detect decreased fat store or loss of subcutaneous fat and signs of muscle wasting. Laboratory parameters are serum albumin and serum total iron binding capacity (TIBC). Each of 10 MIS components is classified among four levels of severity, from 0 (normal) to 3 (severely abnormal). The sum of all 10 MIS components ranges from 0 (normal) to 30 (severely malnourished); a higher score reflects a more severe degree of malnutrition and inflammation.

Definitions of sarcopenia, obesity, and sarcopenic obesity

The investigators determine the presence of sarcopenia according to the European Working Group on Sarcopenia in Older People(EWGSOP) consensus definition. A diagnosis of sarcopenia requires the presence of low muscle mass in addition to a low handgrip strength or a slow gait speed.

Participants were considered to have severe sarcopenia if all three of these criteria were present, whereas those with low muscle mass, but without a low handgrip strength or a slow gait speed, were considered to be in the pre-sarcopenia stage.

Obesity was defined in 3 ways

1. Base on waist circumference:

   waist circumference was measured at the mid-level between the iliac crest and the lower border of the twelfth rib while the subject stood with feet 25-30 cm apart. A normal WC level in men and women was defined as <90 and <80 cm, respectively.
2. Based on the reference values by Baumgartner et al. The cut-off point of obesity was a body fat percentage that is greater than the 60th percentile of the study sample by sex (27.82% in men and 37.61% in women).
3. Based on BMI: The investigators calculate the BMI as the bodyweight in kg divided by the square of the height in m2, and categorized it according to the definition of the Department of Health in Taiwan (BMI 24-26.9 kg/m2 for overweight and BMI ≥27 kg/m2 for obesity).

Sarcopenic obesity is characterized by high body fat combined with low skeletal muscle mass. Class II sarcopenia was indicated by definition in participants whose height- or weight-adjusted ASM was below 2 Standard Deviation(SD). SO was considered as the combination of class II sarcopenia and obesity according to each definition.

Covariates

The covariates were the participant's age, sex, smoking status (smoker or non-smoker), and comorbidities. Participants who reported smoking cigarettes at the time of the interview were defined as smokers. Comorbidities were assessed by referring to the self-reported physician's diagnosis, and included hypertension, cancer, advanced liver disease, diabetes mellitus, stroke, heart failure, arthritis, and chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes aged > 20 years-old.
* Received stable hemodialysis at least 3 months.
* Written informed consent.

Exclusion Criteria:

* Patients with malignant disease, acute infectious disease, acute inflammatory disease,liver cirrhosis, and chronic use of any type of immunosuppressive medication are excluded.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis (HD) patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Presence of sacropenia | one year
  Definition and diagnosis of sarcopenia from European European Working Group on Sarcopenia based on 1. Low muscle mass 2. Low muscle strength 3. Low physical performance

CONTACTS AND LOCATIONS:
Overall Officials: Mei-An Pai, MD, Principal Investigator — Tungs' Taichung Metroharbour Hospital

IPD SHARING:
Plan to Share IPD: Yes